CLINICAL TRIAL: NCT04133298
Title: Evaluation of Tunneling Technique With Subepithelial Connective Tissue Graft Vs. Laser De-epithelialized Gingival Graft in Management of Multiple Cairo RT-2 Gingival Recessions.
Brief Title: Evaluation of SECTG Vs. Laser-DGG in Management of Gingival Recessions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25354999
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: * Blinding of the participants is not applicable.
  * Blinding of the operator is not applicable.
  * The outcome assessor and biostatistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tunneling with laser de-epithelized gingival graft. (Active Comparator): After the administration of local anesthesia, the dimension of the needed graft will be marked by a #15c blade and then diode laser de-epithelization will take place. The de-epithelized area will be then harvested using a # 15c blade. The donor site will be covered by cyanoacrylate tissue adhesive dressing .
  Interventions: Procedure: Tunneling with laser de-epithelized gingival graft
- Tunnelingwith subepithelial connective tissue graft. (Active Comparator): After administration of local anesthesia. A single incision will be made to the bone in a horizontal direction 3mm apical to the gingival margin of the maxillary teeth. The length of the incision will be determined by the dimensions of the graft required. A partial-thickness dissection will be then made within the single incision aiming to harvest an average thickness of two mm subepithelial connective tissue. Then, the graft will be carefully elevated from the palate with the use of the blade. Primary closure will be obtained using 4-0 polyglycolic acid.
  Interventions: Procedure: Tunnelingwith subepithelial connective tissue graf

INTERVENTIONS:
Procedure: Tunneling with laser de-epithelized gingival graft — After the administration of local anesthesia, the dimension of the needed graft will be marked by a #15c blade and then diode laser de-epithelization will take place. The de-epithelized area will be then harvested using a # 15c blade. The donor site will be covered by cyanoacrylate tissue adhesive dressing .
  Arms: Tunneling with laser de-epithelized gingival graft.
Procedure: Tunnelingwith subepithelial connective tissue graf — After administration of local anesthesia. A single incision will be made to the bone in a horizontal direction 3mm apical to the gingival margin of the maxillary teeth. The length of the incision will be determined by the dimensions of the graft required. A partial-thickness dissection will be then made within the single incision aiming to harvest an average thickness of two mm subepithelial connective tissue. Then, the graft will be carefully elevated from the palate with the use of the blade. Primary closure will be obtained using 4-0 polyglycolic acid
  Arms: Tunnelingwith subepithelial connective tissue graft.

SUMMARY:
This study evaluates laser de-epithelialized gingival graft to be as effective as subepithelial connective tissue graft in management of multiple gingival recessions using tunneling technique. half pf participants will be treated from gingival recession using tunneling technique with laser de-epithelized gingival graft, while the other half will be treated using tunneling technique with subepithelial connective tissue graft.

DETAILED DESCRIPTION:
Tunneling technique is a minimal invasive method for coronal advancement during gingival recession coverage. The technique provide better blood supply which enhances wound healing and results in successful root coverage and attachment gain. Tunneling technique is suggested to be incorporated with a soft tissue tissue for better recipient site outcome.

In a systemic review and meta-analysis conducted in 2019 there was limited evidence available comparing subepithelial connective tissue graft to the de-epithelialized gingival graft. However the de-epithelialized gingival graft showed superior mean root coverage, keratinized tissue gain and clinical attachment gain over the subepithelial connective tissue graft making it the technique of choice when incorporated with coronal advancement flap in treatment of gingival recession. Laser de-epithelization may enrich the advantages of the conventional de-epithelization method where more uniform predictable epithelization can be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior teeth and premolars with multiple Miller's Class I and II gingival recessions.
2. Identifiable cemento-enamel junction.
3. The teeth with gingival recessions are vital teeth.
4. Plaque Index and Gingival bleeding index less than 20% after phase one therapy.

Exclusion Criteria:

1. Patients with systemic diseases and medical conditions that may affect the treatment outcomes.
2. Prosthetic crown, restoration or tooth decay involving the CEJ.
3. Previous periodontal surgery in the area of interest.
4. Smokers.
5. Pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Gingival Thickness gain | 6 month
  it will be calculated based on volumetric difference of a defined area located on attached gingiva above the site to be corrected surgically, that is by taking a base line digital impression and superimpose it to another digital impression 6 month postoperatively. Buccal tooth surface will be used as a reference for the superimposition procedure. The digital measurements will be taken to nearest 0.01mm. Finally, gingival thickness gain will be calculated as the measured volume gain per measured area, [Gingival thickness gain (mm) = volume (mm3) / area (mm2)].

SECONDARY OUTCOMES:
root coverage gain | 6 month
  it will be calculated digitally by comparing base line digital impression to a 6 month postsurgical digital impression. A digital ruler will be used to measure the distance from gingival margin to the cemento-enamel junction on a point mid-buccally pre-surgically then post-surgically. The digital measurements will be taken to nearest 0.01mm.
  Mean of root coverage and its percentage will be calculated. Mean root coverage will be measured in millimeters and percentage in percent.
Keratinized tissue width gain | 6 month
  Will be measured by a periodontal probe from the gingival margin to the mucogingival junction, at the mid buccal area.
Probing depth | 6 month
  Will be measured by a periodontal probe from the base of sulcus/pocket to the gingival margin mid- buccally.
Clinical attachment level gain | 6 month
  Will be measured by a periodontal probe from the base of sulcus/pocket to the cement enamel junction mid- buccally.
Post-operative pain score | 2 weeks
  Patients will be questioned in arabic after two weeks post-operative to assess pain, number of analgesic pills taken and number of days pills were taken. That will be assessed by visual analog scale (VAS) graduated from one to ten, where one indicates minimal pain and ten refers to severe pain.
Patient satisfaction | 2 weeks
  Patients will be questioned in arabic about the palatal wound after two weeks of the surgery. The questionnaire will include four graduated visual analog scales to describe pain intensity, hemorrhage intensity, fear of jeopardizing the palatal wound, their chewing ability, their willingness to perform the surgery another time if needed and their satisfaction about the esthetic outcome after the surgery. Graduation will be from one to ten, where one indicates minimal and ten refers to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Akawi, Principal Investigator — Cairo University
Locations (1):
- CairoU, Cairo, Egypt